CLINICAL TRIAL: NCT05624190
Title: Intra-arterial Recombinant Human Tenecteplase Tissue-type Plasminogen Activator rhTNK-tPA) Thrombolysis for Acute Large Vessel Occlusion After Successful Mechanical Thrombectomy Recanalization -- A Multicenter, Prospective, Randomized, Open-label, Blinded End-point Trial (ANGEL-TNK)
Brief Title: Intra-arterial Recombinant Human TNK Tissue-type Plasminogen Activator (rhTNK-tPA) Thrombolysis for Acute Large Vascular Occlusion After Successful Mechanical Thrombectomy Recanalization
Acronym: ANGEL-TNK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director of Department of interventional neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2022041
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TNK group (Experimental): Patients of this group will receive IA rhTNK-tPA plus Best Medical Management (BMM) after successful mechanical thrombectomy (MT) recanalization
  Interventions: Drug: Recombinant Human tenecteplase Tissue-type Plasminogen Activator (rhTNK-tPA); Other: Best Medical Management
- control group (Active Comparator): Patients of this group will receive Best Medical Management (BMM) alone after successful mechanical thrombectomy (MT) recanalization
  Interventions: Other: Best Medical Management

INTERVENTIONS:
Drug: Recombinant Human tenecteplase Tissue-type Plasminogen Activator (rhTNK-tPA) — The administration of rhTNK-tPA will be infused constant and slowly over 15min (0.125 mg/kg, Max 12.5mg) through a microcatheter.
  Other Names: IA rhTNK-tPA
  Arms: TNK group
Other: Best Medical Management — Best Medical Management

SUMMARY:
The goal of this clinical trial is to evaluate whether intra-arterial (IA) rhTNK-tPA thrombolysis can improve neurological outcomes in acute large vessel occlusion patients after successful mechanical thrombectomy (MT) recanalization between 4.5- 24 hours from symptom onset. Participants enrolled will be randomly assigned to study or control arm with a 1:1ratio. Study group will receive IA rhTNK-tPA thrombolysis (0.125 mg/kg, Max 12.5mg) plus best medical management, and control receive best medical management alone.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

1. Age >18 years;
2. NIHSS ≥2;
3. Onset of symptoms to baseline CT imaging time: 4.5 to 24 hours, including wake-up stroke and unwitnessed stroke; Time of onset of symptoms is defined as "last known well" (LKW);
4. Pre-stroke mRS score 0-1;
5. Signed informed consent from patient or their health care proxy.

Neuroimaging Inclusion Criteria:

1. CTA/MRA proven intracranial artery occlusion: Intracranial Internal Carotid Artery (ICA)、M1 of Middle cerebral artery (MCA)、dominant M2 of MCA;
2. ASPECTS ≥6 on non-contrast CT (NCCT) scan or DWI MRI;
3. CT perfusion or MR perfusion: ischemic infarct core <70ml, mismatch ratio≥1.2, mismatch volume ≥15ml;
4. Treated with MT resulting in an eTICI score 2b50-3 at end of the procedure. Patients with an eTICI score 2b50-3 on the diagnostic cerebral angiography before the onset of MT are also eligible for the study.

Exclusion Criteria:

Clinical Exclusion Criteria:

1. IV thrombolysis used on admission;
2. Contraindications to intravenous thrombolysis;
3. Balloon angioplasty, permanent stenting and other situations during the endovascular procedure that require antiplatelet therapy or anticoagulant within the first 24h;
4. IV heparin (heparinized saline allowed);
5. Females who are pregnant, or those of child-bearing potential with positive urine or serum beta Human Chorionic Gonadotropin (HCG) test;
6. Brain tumor (with mass effect);
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
8. Known coagulopathy, INR>1.7 or use of novel anticoagulants < 48h from symptom onset
9. Platelets < 50*109/L;
10. Suspicion of septic emboli or endocarditis
11. Renal Failure as defined by a serum creatinine > 2.5 mg/dl (or 220μmol/l) or glomerular Filtration Rate [GFR] < 30ml/min;
12. Patient who requires hemodialysis or peritoneal dialysis, or who has a contraindication to angiogram for whatever reason;
13. Suspicion of aortic dissection;
14. Parenchymal organ surgery and biopsy were performed in the past one month;
15. Any active bleeding or recent bleeding (gastrointestinal bleeding, urinary bleeding, etc.) in the past 1 month;
16. History of life-threatening allergy (more than rash) to contrast medium;
17. SBP >185 mmHg or DBP >110 mmHg refractory to treatment;
18. Serious, advanced, terminal illness with anticipated life expectancy < 6 months;
19. Participation in another randomized clinical trial that could confound the evaluation of the study;
20. Other circumstances that the investigator considers inappropriate for participation or may pose a significant risk to patients (e.g. inability to understand and/or comply with study procedures and/or follow-up due to mental disorders, cognitive or mood disorders).

Specific Neuroimaging Exclusion Criteria

1. Midline shift or herniation, mass effect with effacement of the ventricles
2. Evidence of acute intracranial hemorrhage on CT/MRI
3. Acute bilateral strokes or multiple intracranial vessel occlusions
4. Isolated extracranial ICA occlusion or tandem carotid / MCA occlusion
5. Dissection of occluded artery on DSA after thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Rate of excellent outcome | 90±7 days after randomization
  Rate of 90 (±7) day modified Rankin scale (mRS) 0-1

SECONDARY OUTCOMES:
Rate of sICH (Heidelberg Bleeding Classification) | within 48 hours after randomization
  Rate of sICH (Heidelberg Bleeding Classification)
Volume of Tmax>6s | 24 hours (±12 hours) after randomization
Infarct core volume change from baseline | 7 days (±1 day) after randomization/at discharge or at 36 hours (±12 hours) after randomization
  Infarct core volume change from baseline, assessed with NCCT at 7 days (±1 day) after randomization/at discharge or with MRI at 36 hours (±12 hours)
mRS (shift analysis) | 90 days (±7 days) after randomization
  mRS (shift analysis)
Rate of good outcome | 90 days (±7 days) after randomization
  Rate of mRS 0-2
Rate of mRS 0-3 | 90 days (±7 days) after randomization
  Rate of mRS 0-3
NIHSS 0-1 or decrease ≥10 from baseline NIHSS | 36 hours (±12hours) after randomization
  NIHSS 0-1 or decrease ≥10 from baseline NIHSS
EQ-5D-5L score | 90 days (±7 days) after randomization
  EQ-5D-5L score
All-caused mortality | 90 days (±7 days) after randomization
  All-caused mortality
Rate of any intracranial hemorrhage (Heidelberg Bleeding Classification) | within 48 hours after randomization
  Rate of any intracranial hemorrhage (Heidelberg Bleeding Classification)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Miao Z, Luo G, Song L, Sun D, Chen W, Yao X, Pan Y, Liu Y, Yuan G, Wen C, Wei M, Cai X, Yang Q, Zhou Z, Chang M, Nan G, Wang J, Xiang G, Zhou L, Gao W, Zhang H, Hao J, Xu C, Sun Y, Yi T, Feng G, Han H, Gao F, Ma N, Mo D, Sun X, Deng Y, Tong X, Li X, Jia B, Wang B, He Z, Yang M, Zhao X, Zhang X, Zhang L, Li S, Tong X, Jing J, Xiong Y, Liu T, Li Z, Ren Z, Wang Y, Liebeskind DS, Jovin TG, Nguyen TN, Wang Y, Liu L, Yan B, Huo X; ANGEL-TNK Investigators. Intra-arterial Tenecteplase for Acute Stroke After Successful Endovascular Therapy: The ANGEL-TNK Randomized Clinical Trial. JAMA. 2025 Aug 19;334(7):582-591. doi: 10.1001/jama.2025.10800. PMID 40616323
- [Derived] Huo X, Luo G, Sun D, Nguyen T, Abdalkader M, Chen W, Yao X, Yuan G, Yi T, Han H, Pan Y, Jovin TG, Liebeskind DS, Liu L, Zhao X, Ren Z, Wang Y, Wang Y, Yan B, Miao Z. Intra-arterial tenecteplase after successful endovascular therapy (ANGEL-TNK): protocol of a multicentre, open-label, blinded end-point, prospective, randomised trial. Stroke Vasc Neurol. 2025 Aug 26;10(4):508-513. doi: 10.1136/svn-2024-003318. PMID 39357896